CLINICAL TRIAL: NCT02874365
Title: Intestinal Stem Cells Characterization in Intestinal Organoid Culture From Inflammatory Bowel Disease and Intestinal Polyposis Patients
Brief Title: Intestinal Stem Cells Characterization
Acronym: BIODIGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/15/7816
Record Dates: First submitted 2016-05-13; First posted 2016-08-22 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Crohn disorder (Experimental): arm composed by 30 patients with Crohn disorder
  Interventions: Procedure: Endoscopic biopsies
- FAP (familial adenomatous polyposis ) (Experimental): arm composed by 30 patients with FAP disorder
  Interventions: Procedure: Endoscopic biopsies
- ulcerative colitis (Experimental): arm composed by 30 patients with ulcerative colitis
  Interventions: Procedure: Endoscopic biopsies
- witness (Sham Comparator): arm composed by 30 patients with no intestinal disorders
  Interventions: Procedure: Endoscopic biopsies

INTERVENTIONS:
Procedure: Endoscopic biopsies — intestinal biopsies

SUMMARY:
A monocentric pilot studying intestinal organoids from endoscopic biopsies of IBD (Crohn and ulcerative colitis), FAP patients and healthy controls. Investigate the morphological characteristics of organoids, the expression of genes and proteins of the Wnt/APC/beta-catenin pathway within both ISC.

DETAILED DESCRIPTION:
Intestinal organoids are 3D mini-guts produced in vitro based on intestinal stem cell (ISC) capabilities. These organoids contain all of the intestinal epithelial cells. The renewal of the two kinds of ISCs, which are present at the bottom of intestinal crypts, is controlled by Wnt/APC/beta-catenin pathway. Mutations of genes involved in this pathway are found in intestinal polyposes like familial adenomatous polyposis (FAP, APC gene).

This model is of interest to study early pathophysiological events occurring within intestinal epithelium, in the context of FAP and inflammatory bowel diseases (IBD). An excessive proliferation or an abnormal healing is found in FAP and IBD respectively. Investigators hypothesized that it could specifically involved one of the 2 ISCs. Columnar basal cells (CBC) and ISC located at the +4 position from the bottom of the crypt (ISC+4) can both differentiate into absorptive or secretory intestinal epithelial cells. However, CBC and ISC+4 could have different metabolic, migratory functions, or stress survival.

Investigators designed a monocentric pilot study to develop intestinal organoids from endoscopic biopsies of IBD (Crohn and ulcerative colitis), FAP patients and healthy controls. Investigators plan to investigate the morphological characteristics of organoids, the expression of genes and proteins of the Wnt/APC/beta-catenin pathway within both ISC. Will also be studied the expression of key genes of tumor initiation (PTEN, BMPR1A, p53 and KRAS) and inflammatory parameters (cytokines and lipid mediators).

The results of this study could improve the understanding of intestine renewal. Later on, the development of new drugs could beneficiate to IBD and FAP patients.

ELIGIBILITY:
Inclusion Criteria: patient must have a coloscopy for intestinal pain -

Exclusion Criteria: cancer

-

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-09; Primary Completion 2022-12 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
number of organoids | 2 days
  number of organoids in culture wells during the follow-up

SECONDARY OUTCOMES:
mean size of organoids | 2 days
  mean diameter of organoids in culture wells during the follow-up
percentage of different types of organoids | 2 days
  organoids are differentiated by the size of the epithelial cell border and by the presence or absence of buds

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MAS, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hopital des Enfants, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laborde N, Barusseaud A, Quaranta M, Rolland C, Arrouy A, Bonnet D, Kirzin S, Sola-Tapias N, Hamel D, Barange K, Duffas JP, Gratacap MP, Guillermet-Guibert J, Breton A, Vergnolle N, Alric L, Ferrand A, Barreau F, Racaud-Sultan C, Mas E. Human colonic organoids for understanding early events of familial adenomatous polyposis pathogenesis. J Pathol. 2025 Jan;265(1):26-40. doi: 10.1002/path.6366. Epub 2024 Dec 6. PMID 39641466
- [Background] Moreau J, Mas E. Drug resistance in inflammatory bowel diseases. Curr Opin Pharmacol. 2015 Dec;25:56-61. doi: 10.1016/j.coph.2015.11.003. Epub 2015 Nov 29. PMID 26645664